CLINICAL TRIAL: NCT05886322
Title: Comparison of Patient Reported Disease Activity Scores Combined With Fecal Calprotectin Home Tests for Remote Monitoring of IBD Patients: a Multicenter Prospective Validation Study
Brief Title: Remote Monitoring of IBD
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Maastricht University Medical Center (Other)
Collaborators: Maastricht University (Other)
Responsible Party: Sponsor
Other Study IDs: NL75205.068.20; NL9313 (Registry Identifier: Netherlands Trial Register)
Record Dates: First submitted 2023-04-26; First posted 2023-06-02 (Actual); Last update posted 2023-06-02 (Actual); Status verified 2023-05

CONDITIONS: Inflammatory Bowel Diseases; Crohn Disease; Ulcerative Colitis
Keywords: fecal calprotectin; patient reported outcome measures; mucosal inflammation
MeSH Terms: conditions — Inflammatory Bowel Diseases; Crohn Disease; Colitis, Ulcerative; Mucositis | interventions — Colonoscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: patient reported outcome measures — MIAH, mHI, Manotiba IBD Index, p-HBI/SCCAI, IBD-control
Diagnostic Test: fecal calprotectin — fecal calprotectin point-of-care test and laboratory test
Diagnostic Test: colonoscopy — endoscopic activity scores (SES-CD, UCEIS, MES)

SUMMARY:
Crohn's disease (CD) and ulcerative colitis (UC) are chronic inflammatory bowel diseases (IBD) with a heterogeneous disease course. Recurrent mucosal inflammation or chronic subclinical inflammation results in damage to the bowel and complications like stenosis, fistula and colorectal cancer. Therefore, tight control of mucosal inflammation is important to prevent complications.

The goal of this multicenter observational cohort study is to determine the best remote monitoring tool for predicting mucosal inflammation in adult patients with inflammatory bowel disease, relative to the gold standard endoscopy.

Participants will be asked to fill out questionnaires regarding disease activity (MIAH, mHI, IBD-control, Manitoba IBD Index, p-HBI/p-SCCAI), perform a FC home test and collect one stool sample for routine laboratory calprotectin measurement, before the start of the bowel preparation for the ileocolonoscopy. During this ileocolonoscopy, endoscopic disease activity will be determined.

.

ELIGIBILITY:
Inclusion Criteria:

* Established diagnosis of CD or UC according to ECCO guidelines
* CD or UC patients scheduled for an ileocolonoscopy, or UC patients scheduled for an sigmoidoscopy at the endoscopy ward of one of the participating centers (regardless of indication)
* Aged 18 years or older
* Smartphone with internet access (for use FC home test)

Exclusion Criteria:

* Unclassified IBD
* Ileostomy, colostomy, ileoanal pouch anastomosis or ileorectal anastomosis
* Isolated upper gastro-intestinal CD, or isolated peri-anal disease
* Insufficient knowledge of Dutch language

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with an established diagnosis of CD or UC, scheduled for an ileocolonoscopy or sigmoidoscopy as part of routine care at the endoscopy ward of one of the participating centers, are eligible for participation.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2022-06-07 (Actual); Primary Completion 2024-06 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Prediction of mucosal inflammation in daily clinical practice with PROMs and FC home test | week 0 (i.e. in the week before the colonoscopy)
Recalibration of PROMs | week 0 (i.e. in the week before the colonoscopy)
  Recalibrate PROMs with the FC home test to optimise prediction of mucosal inflammation, relative to the gold standard ileocolonoscopy, for use in daily clinical practice

SECONDARY OUTCOMES:
prediction of mucosal inflammation in strict trial setting with PROMs and FC home test | week 0 (i.e. in the week before the colonoscopy)
Agreement between FC home test and routine laboratory tests | week 0-1 (i.e. FC home test in the week before the colonoscopy and the laboratory test at the day of the colonoscopy)
Association between clinical (abdominal pain) and histologic disease activity | week 0-1
Association between IBD-control and histologic disease activity | week 0-1

CONTACTS AND LOCATIONS:
Overall Officials: prof. dr. Pierik, Principal Investigator — Maastricht University Medical Centre
Locations (5):
- Netherlands (5):
  - Jeroen Bosch Hospital, 's-Hertogenbosch
  - Catharina Hospital Eindhoven, Eindhoven
  - Maastricht University Medical Centre, Maastricht
  - Franciscus Gasthuis&Vlietland, Rotterdam
  - Zuyderland Medical Centre, Sittard

REFERENCES:
- [Background] de Jong MJ, Roosen D, Degens JHRJ, van den Heuvel TRA, Romberg-Camps M, Hameeteman W, Bodelier AGL, Romanko I, Lukas M, Winkens B, Markus T, Masclee AAM, van Tubergen A, Jonkers DMAE, Pierik MJ. Development and Validation of a Patient-reported Score to Screen for Mucosal Inflammation in Inflammatory Bowel Disease. J Crohns Colitis. 2019 Apr 26;13(5):555-563. doi: 10.1093/ecco-jcc/jjy196. PMID 30476099
- [Background] Van Deen WK, van der Meulen-de Jong AE, Parekh NK, Kane E, Zand A, DiNicola CA, Hall L, Inserra EK, Choi JM, Ha CY, Esrailian E, van Oijen MG, Hommes DW. Development and Validation of an Inflammatory Bowel Diseases Monitoring Index for Use With Mobile Health Technologies. Clin Gastroenterol Hepatol. 2016 Dec;14(12):1742-1750.e7. doi: 10.1016/j.cgh.2015.10.035. Epub 2015 Nov 18. PMID 26598228
- [Background] Bennebroek Evertsz' F, Hoeks CC, Nieuwkerk PT, Stokkers PC, Ponsioen CY, Bockting CL, Sanderman R, Sprangers MA. Development of the patient Harvey Bradshaw index and a comparison with a clinician-based Harvey Bradshaw index assessment of Crohn's disease activity. J Clin Gastroenterol. 2013 Nov-Dec;47(10):850-6. doi: 10.1097/MCG.0b013e31828b2196. PMID 23632348
- [Background] Bennebroek Evertsz' F, Nieuwkerk PT, Stokkers PC, Ponsioen CY, Bockting CL, Sanderman R, Sprangers MA. The patient simple clinical colitis activity index (P-SCCAI) can detect ulcerative colitis (UC) disease activity in remission: a comparison of the P-SCCAI with clinician-based SCCAI and biological markers. J Crohns Colitis. 2013 Dec;7(11):890-900. doi: 10.1016/j.crohns.2012.11.007. Epub 2012 Dec 24. PMID 23269224
- [Background] Bodger K, Ormerod C, Shackcloth D, Harrison M; IBD Control Collaborative. Development and validation of a rapid, generic measure of disease control from the patient's perspective: the IBD-control questionnaire. Gut. 2014 Jul;63(7):1092-102. doi: 10.1136/gutjnl-2013-305600. Epub 2013 Oct 9. PMID 24107590
- [Background] Clara I, Lix LM, Walker JR, Graff LA, Miller N, Rogala L, Rawsthorne P, Bernstein CN. The Manitoba IBD Index: evidence for a new and simple indicator of IBD activity. Am J Gastroenterol. 2009 Jul;104(7):1754-63. doi: 10.1038/ajg.2009.197. Epub 2009 May 19. PMID 19455122
- [Derived] Janssen L, van Linschoten RCA, West RL, Gilissen LPL, Romberg-Camps M, Brandts L, Mujagic Z, Romkens TE, Pierik M. Predicting mucosal inflammation in IBD patients using patient-reported symptom scores and a faecal calprotectin home test: protocol for a multicentre prospective validation study. BMJ Open. 2024 Oct 7;14(10):e076290. doi: 10.1136/bmjopen-2023-076290. PMID 39375184